CLINICAL TRIAL: NCT04560387
Title: Effect of Complex Weight-reducing Interventions on Rhythm Control in Obese Subjects With Atrial Fibrillation
Acronym: HOBIT-FS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Martin Haluzik (Other Government)
Responsible Party: Sponsor-Investigator, Martin Haluzik, Prof. Martin Haluzik, DSc., Institute for Clinical and Experimental Medicine
Organization: Institute for Clinical and Experimental Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NU20-02-00190
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Atrial Fibrillation; Obesity
MeSH Terms: conditions — Atrial Fibrillation; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Physician-lead complex program of weight-reducing interventions including education, diet counselling and regular physical activity aimed at achieving and maintaining a 10% reduction of baseline body weight.
  Bariatric surgery - sleeve gastrectomy in a subgroup of subjects with BMI > 35 kg/m2, i.e. standard indication of bariatric surgery (patients with BMI > 35 kg/m2 and a presence of metabolic or other complications).
  Interventions: Behavioral: Physician-lead complex program of weight-reducing interventions; Procedure: Bariatric surgery - sleeve gastrectomy
- Conservative (No Intervention): Routine treatment of obesity

INTERVENTIONS:
Behavioral: Physician-lead complex program of weight-reducing interventions — A structured motivational and goal directed program will be used for weight reduction involving physicians, nutritionists, educators and physiotherapists. Initially, based on the input data provided by the patient an individual nutritional plan will be designed with the aim of reducing caloric intake by 10%. Low-intensity aerobic exercise for 30 min will be prescribed 3-times a week with the aim of increasing the frequency to 5-times a week and participants will be offered the possibility to participate in regular physiotherapist-lead group exercises. Patients will be required to maintain a diet and physical activity diary. Regular reviews will be scheduled every 3-6 months according to the actual weight loss.
  Arms: Interventional
Procedure: Bariatric surgery - sleeve gastrectomy — Bariatric surgery will be performed based on actual medical indication and independently of patient's participation in the study. Sleeve gastrectomy was selected as the currently most frequent restrictive type of bariatric surgery with a proven efficacy on weight reduction, metabolic status and low-grade inflammation
  Arms: Interventional

SUMMARY:
Obesity is a well-established risk factor for the development of atrial fibrillation (AF), while the reduction of body weight was shown to reduce the risk of AF. However, little is known about the effect of different weight-reducing interventions on AF burden. The study will evaluate the effect of a complex program aimed at weight reduction on AF burden in subjects after catheter ablation for AF and at least 1st degree obesity. This will be investigated in randomized study design and compared with patients receiving standard care without specific obesity-related intervention. The weight loss program will consist of diet, lifestyle and exercise counselling and, in selected subjects, also bariatric surgery in order to achieve a sustained weight loss of >10% of initial body weight. Secondary aims include identification of patient phenotypes with the most benefits from weight reduction as well as elucidation of potential pathomechanisms linking obesity and AF, with the main focus being on low-grade inflammation. The project will help to define the optimal weight-reducing regimen in AF and to tailor the interventions to individual patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent AF scheduled for primary RF ablation
* BMI ≥30 kg/m2
* Age 18-70 years
* Informed consent to the study

Exclusion Criteria:

* Previous ablation for AF
* Myocardial infarction, stroke or pulmonary embolism < 3 months prior to inclusion
* left ventricular ejection fraction < 40%
* Left atrium diameter > 55 mm
* Active thyroid disease
* Chronic kidney disease stage IV-V (eGFR < 0.5 ml/s)
* Chronic liver disease
* Active malignancy
* Inability to comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | 18 months
  Atrial fibrillation burden expressed as % of total monitoring time at final visit

SECONDARY OUTCOMES:
Number of AF episodes on 14-day Holter monitoring | 18 months
  Number of AF episodes on 14-day Holter monitoring
Progressive reduction of AF burden between 12- and 18-month follow up visit | 18 months
  Progressive reduction of AF burden between 12- and 18-month follow up visit
hsCRP | 18 months
Epicardial adipose tissue volume | 18 months
  Assessed by transthoracic echocardiography
Concentration of atrial natriuretic peptide (ANP) | 18 months
Concentration of brain natriuretic peptide (BNP) | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Stolbova K, Novodvorsky P, Jakubikova I, Dvorakova I, Mraz M, Wichterle D, Kautzner J, Haluzik M. Effect of Complex Weight-Reducing Interventions on Rhythm Control in Obese Individuals with Atrial Fibrillation Following Catheter Ablation: A Study Protocol. Adv Ther. 2021 Apr;38(4):2007-2016. doi: 10.1007/s12325-021-01667-0. Epub 2021 Mar 12. PMID 33710588